CLINICAL TRIAL: NCT00476281
Title: Multicenter Prospective Study of Abnormalies Tolerance Glucose by the Continuous Measurement of Glucose of Nutritional Status and Breathing in the Patient With Cystic Fibrosis
Brief Title: Nutritional, Metabolic and Respiratory Status in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Association d'Aide aux Insuffisants Respiratoires d'Alsace Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3887
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis; Diabetes
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

ARMS (1):
- abnormal glucose tolerance (Other): abnormal glucose tolerance
  Interventions: Procedure: Urinary collect; Procedure: Continuous Glucose Monitoring System (CGMS)

INTERVENTIONS:
Procedure: Urinary collect
Procedure: Continuous Glucose Monitoring System (CGMS)

SUMMARY:
Diabetes is a important complication of cystic fibrosis (CF). The improved life expectancy of patients with cystic fibrosis, as a result of advances in medical therapy, has resulted in an increasing prevalence of cystic fibrosis-related diabetes (CFRD). CFRD is associated with accelerated pulmonary decline and increased mortality. Pulmonary effects are seen some years before the diagnosis of CFRD implying that impaired glucose tolerance may be very early detrimental. Insulin treatment is clearly indicated in patients with CFRD to control symptoms and reduce complications. However, at the state of impaired glucose tolerance or fasting hyperglycaemia, current screening methods are not suitable for the early management of hyperglycaemia.The recent introduction of the continuous glucose monitoring system (CGMS), which provides a continuous glucose profile, has revealed to be clinically relevant in the investigation of glucose excursions over a long period. This device, widely use in diabetic non cystic fibrosis patients, has been validated in non diabetic cystic fibrosis subjects. Previous studies of continuous glucose monitoring have been realized in CF patients with normal glucose tolerance and diabetes and compared with non CF controlThe aim of our study is to evaluate the glucose profile with continuous glucose monitoring the nutritional and respiratory status in cystic fibrosis subjects, according to their glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* patients 10 years and older with cystic fibrosis
* not known diabetics with fasting blood glucose <1.26 g / l
* outside periods of exacerbation and / or glucocorticoid therapy
* affiliated to a social security scheme
* having received the results of the mandatory medical examination
* having signed an informed consent

Exclusion Criteria:

* Patient transplanted lung and / or liver
* Subject during participation in an interventional clinical trial
* unable to give informed about the information
* patient under judicial protection
* patient under tutorship or curatorship
* pregnancy
* breastfeeding
* patient treated with the combination lumacaftor and ivacaftor

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-04; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
nutritional and respiratory parameters | five years
  descriptive comparison of nutritional and respiratory parameters in function abnormalities glucose tolerance.

SECONDARY OUTCOMES:
abnormal glucose tolerance | five tears
  assess the prevalence of abnormal glucose tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence KESSLER, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (9):
- France (9):
  - Centre Robert Debré - CHU Angers, Angers
  - Service d'Endocrinologie et Métabolisme - CHRU de Lille, Lille
  - Hôpital Laennec - CHU de Nantes, Nantes
  - Service de Pédiatrie A - CHU de Reims, Reims
  - CRCM Centre de Perharidy, Roscoff
  - Service d'Endocrinologie, Diabète et Maladies Métaboliques - Hôpital Civil, Strasbourg
  - Service de Réanimation Médicale - Hôpital Civil, Strasbourg
  - Service de Pneumologie - Hôpital de Hautepierre, Strasbourg
  - Service de Pédiatrie II, Strasbourg

REFERENCES:
- [Derived] Leclercq A, Gauthier B, Rosner V, Weiss L, Moreau F, Constantinescu AA, Kessler R, Kessler L. Early assessment of glucose abnormalities during continuous glucose monitoring associated with lung function impairment in cystic fibrosis patients. J Cyst Fibros. 2014 Jul;13(4):478-84. doi: 10.1016/j.jcf.2013.11.005. Epub 2013 Dec 17. PMID 24359972